CLINICAL TRIAL: NCT04837547
Title: PEACH TRIAL- Precision mEdicine and Adoptive Cellular tHerapy for the Treatment of Recurrent Neuroblastoma and Newly Diagnosed Diffuse Intrinsic Pontine Glioma (DIPG)
Brief Title: PEACH TRIAL- Precision Medicine and Adoptive Cellular Therapy
Acronym: PEACH
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Beat Childhood Cancer Research Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCC017
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Neuroblastoma; Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Neuroblastoma; Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Subjects with Diffuse Intrinsic Pontine Glioma (DIPG). (Experimental): This Phase I study is will utilize a standard 3+3 dose escalation design to establish the MTD and will evaluate the following three pre-specified dose levels of xALT:
  Dose Level 1: 3 x10^7 cells/kg Dose Level +1: 3 x10^8 cells/kg Dose Level -1: 3 x10^6 cells/kg
  The dose escalation scheme will be evaluated for Arm 1 and Arm 2 separately. For each Study Arm, a minimum of 4 DLT evaluable subjects and a maximum of 12 DLT evaluable subjects will be enrolled (a total of 8 to 24 DLT evaluable subjects).
  Interventions: Biological: Tumor-specific ex vivo expanded autologous lymphocyte transfer (TTRNA-xALT)
- Arm 2: Relapsed/Refractory Neuroblastoma (NB) (Experimental): This Phase I study is will utilize a standard 3+3 dose escalation design to establish the MTD and will evaluate the following three pre-specified dose levels of xALT:
  Dose Level 1: 3 x10^7 cells/kg Dose Level +1: 3 x10^8 cells/kg Dose Level -1: 3 x10^6 cells/kg
  The dose escalation scheme will be evaluated for Arm 1 and Arm 2 separately. For each Study Arm, a minimum of 4 DLT evaluable subjects and a maximum of 12 DLT evaluable subjects will be enrolled (a total of 8 to 24 DLT evaluable subjects).
  Interventions: Biological: Tumor-specific ex vivo expanded autologous lymphocyte transfer (TTRNA-xALT)

INTERVENTIONS:
Biological: Tumor-specific ex vivo expanded autologous lymphocyte transfer (TTRNA-xALT) — There will be two immunotherapy products manufactured and administered to subjects enrolled on this trial. The first product will be autologous dendritic cells (DCs) loaded with total tumor messenger ribonucleic acid (mRNA) (TTRNA) derived from malignant tumors. The second product will be autologous T lymphocytes stimulated ex vivo against TTRNA antigens for autologous transfer (TTRNA-xALT). DCs are professional antigen-presenting cells critical for the initiation of B and T-cell responses in vivo.
  Other Names: xALT

SUMMARY:
A Phase I open-label, multicenter study, to evaluate the safety, feasibility, and maximum tolerated dose (MTD) of treating children with newly diagnosed DIPG or recurrent neuroblastoma with molecular targeted therapy in combination with adoptive cell therapy (Total tumor mRNA-pulsed autologous Dendritic Cells (DCs) (TTRNA-DCs), Tumor-specific ex vivo expanded autologous lymphocyte transfer (TTRNA-xALT) and Autologous G-CSF mobilized Hematopoietic Stem Cells (HSCs)).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have proven pediatric cancer with confirmation at diagnosis or at the time of recurrence/progression and clinical determination of disease for which there is no known effective curative therapy or disease that is refractory to established proven therapies fitting into one of the following categories:
* Disease Status:

High Risk Neuroblastoma-

1. Patients that have relapsed following standard of care therapy or having progressed during standard of care therapy and non-responsive/progressive to accepted curative chemotherapy.
2. Neuroblastoma must be age >12 months at enrollment

Diffuse Intrinsic Pontine (or other brain stem) Glioma

1. Newly-diagnosed patients willing to undergo biopsy
2. Must be within 2 months of diagnosis and prior to starting radiation
3. DIPG must be ≥ 3 years of age at enrollment

   * All subjects must be age ≤ 30 years at enrollment
   * Patient and/or parents/guardian willing to consent to biopsy for obtaining tumor material for confirmatory diagnosis and/or tumor RNA extraction and amplification.
   * Subjects must have measurable disease as defined Per section 8 at the time of biopsy and tumor must be accessible for biopsy. Tumor samples submitted for analysis must contain >30% viable tumor tissue to qualify. In addition, subjects with NB disease confined to the bone marrow are eligible to enroll if the degree of marrow involvement is expected to be >30%.
   * Current disease state must be one for which there is currently no known effective therapy
   * Specimens will be obtained only in a non-significant risk manner and not solely for the purpose of investigational testing.
   * Lansky or Karnofsky Score must be ≥ 60
   * Bone Marrow:

     1. ANC (Absolute neutrophil count) ≥ 1000/µl (unsupported)
     2. Platelets ≥ 100,000/µl (can be transfused)
     3. Hemoglobin > 8 g/dL (can be transfused)
   * Renal: Serum creatinine ≤ upper limit of institutional normal.
   * Adequate liver function must be demonstrated, defined as:

     1. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age AND
     2. ALT (SGPT) ≤ 3 times upper limit of normal (ULN) for age
     3. AST (SGOT) ≤ 3 times upper limit of normal (ULN) for age.
   * Subjects with CNS disease currently taking steroids must have been on a stable dose of steroids for at least one week prior to their biopsy and must not have progressive hydrocephalus at enrollment.
   * A negative serum pregnancy test is required for female participants of childbearing potential (≥13 years of age or after onset of menses)
   * Both male and female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for six months after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrel implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended.
   * Informed Consent: All subjects and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines
   * Post-Biopsy: Patients with post-biopsy neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration.

Exclusion Criteria:

* Absence of tumor on biopsy specimen or a diagnosis other than NBL or glioma on biopsy
* Known autoimmune or immunosuppressive disease or human immunodeficiency virus infection.
* Subjects with significant renal, cardiac, pulmonary, hepatic or other organ dysfunction.
* Prior allergic reaction to GM-CSF or Td.
* Subjects who have received any cytotoxic chemotherapy within the last 7 days prior to biopsy or focal radiotherapy in the case of patients with diffuse intrinsic pontine (or other brain stem) gliomas
* Subjects with NBL who have received any radiotherapy to the primary sample site within the last 14 days (radiation may be included in treatment decision after biopsy).
* Subjects receiving any investigational drug concurrently.
* Subjects with uncontrolled serious infections or a life-threatening illness (unrelated to tumor)
* Subjects with any other medical condition, including malabsorption syndromes, mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the interpretation of the results or which would interfere with a subject's ability to sign or the legal guardian's ability to sign the informed consent, and subject's ability to cooperate and participate in the study

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities as a Measure of Safety and Tolerability | 2 years
  To evaluate the dose-limiting toxicities (DLTs) and to establish the maximum tolerated dose (MTD) of treating children with molecular targeted therapy in combination with adoptive cellular therapy

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years plus 30 days
  To evaluate the overall safety profile of study treatment
Number of Participants that are able to have vaccine produced and delivered | 2 years
  To evaluable the feasibility of producing and administering the protocol directed therapy
Number of participants with progression free survival (PFS) during study | 7 years
  To determine the activity of treatments chosen based on Progression free survival (PFS)
Number of participants with overall survival (OS) during study | 7 years
  To determine the activity of treatments chosen based on Overall Survival (OS)
Determine the Overall Response Rate (ORR) of Participants using INSS Response Evaluation Criteria for NB and RANO criteria for DIPG | 2 years
  To determine the activity of treatments chosen based on Overall Response Rate (ORR)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer at Penn State University; Duane Mitchell, M.D., Ph.D., Study Chair — University of Florida
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Levine Children's Hospital, Charlotte, North Carolina
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Beat Childhood Cancer Consortium website — https://research.beatcc.org/